CLINICAL TRIAL: NCT05852561
Title: Comparison of Combined Superficial and Deep Serratus Anterior Plan Block Versus Deep Serratus Anterior Plan Block for Postoperative Pain Control in Video-Assisted Thoracic Surgery
Brief Title: Comparison of Superficial+Deep Vs. Deep Serratus Anterior Plan Block in Video-Assisted Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Elif Oral Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ataunivatsanalgesia
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Superficial+Deep Serratus Anterior Plan Block (Active Comparator): Superficial+Deep Serratus Anterior Plan Block after Video-Assisted Thoracic Surgery
  Interventions: Other: Group Superficial+Deep Serratus Anterior Plan Block
- Group Deep Serratus Anterior Plan Block (Active Comparator): Deep Serratus Anterior Plan Block after Video-Assisted Thoracic Surgery
  Interventions: Other: Group Deep Serratus Anterior Plan Block

INTERVENTIONS:
Other: Group Superficial+Deep Serratus Anterior Plan Block — The block will be performed after induction of general anesthesia and surgical positioning. 15 ml of 0.375% Bupivacaine + epinephrine 5 µg/ml will be administered between the serratus anterior and latissimus dorsalis muscles. The same concentration of block fluid will be applied between the serratus anterior and the outer intercostal muscle.
  Arms: Group Superficial+Deep Serratus Anterior Plan Block
Other: Group Deep Serratus Anterior Plan Block — 30 ml 0.375% Bupivacaine + epinephrine 5 µg/ml will be administered between the serratus anterior and outer intercostal muscle.
  Arms: Group Deep Serratus Anterior Plan Block

SUMMARY:
Thoracotomy is one of the most painful surgeries; Video-assisted thoracoscopic surgery (VATS) has been developed to reduce the surgical stress of thoracotomy. However, patients may experience moderate to severe pain within the first 24 hours after VATS. Intravenous opioids are frequently used to provide postoperative analgesia, and accordingly, side effects such as postoperative nausea/vomiting and respiratory depression can be seen.

The aim of this study is to compare Superficial+Deep Vs. Deep Serratus Anterior Plan Block for postoperative pain control in VATS cases.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologist's physiologic state I-III patients
2. To undergo Video Assisted Thoracic Surgery
3. Being between the ages of 18-65 years

Exclusion Criteria:

* having a known heart, kidney, liver or hematological disease
* having a history of peptic ulcer, gastrointestinal bleeding, allergy, chronic pain
* Routine analgesic use and history of analgesic use in the last 24 hours
* Not willingto participate in the study
* Uncooperative patients who have coagulopathy or use anticoagulant drugs
* To be allergic to one of the drugs to be used
* Contraindication for Video Assisted Thoracic Surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | first 24 hours
  First 24 hours total fentanyl consumption with patient controlled analgesia

SECONDARY OUTCOMES:
Visual analog pain score | first 48 hours
  Post operative pain will be evaluated with a Visual Analogue Scale (between 0-10; 0: no pain, 10:worst pain) score

CONTACTS AND LOCATIONS:
Overall Officials: Elif Oral Ahiskalioglu, Study Director — Ataturk University
Locations (1):
- Ali Ahiskalioglu, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee J, Kim S. The effects of ultrasound-guided serratus plane block, in combination with general anesthesia, on intraoperative opioid consumption, emergence time, and hemodynamic stability during video-assisted thoracoscopic lobectomy: A randomized prospective study. Medicine (Baltimore). 2019 May;98(18):e15385. doi: 10.1097/MD.0000000000015385. PMID 31045789
- [Background] Qiu L, Bu X, Shen J, Li M, Yang L, Xu Q, Chen Y, Yang J. Observation of the analgesic effect of superficial or deep anterior serratus plane block on patients undergoing thoracoscopic lobectomy. Medicine (Baltimore). 2021 Jan 22;100(3):e24352. doi: 10.1097/MD.0000000000024352. PMID 33546068